CLINICAL TRIAL: NCT00076063
Title: A Phase I/II Clinical Trial to Evaluate the Safety and Immunogenicity of LIPO-5 Alone, ALVAC-HIV (vCP1452) Alone, and ALVAC Prime/LIPO-5 Boost in Healthy, HIV-1 Uninfected Adult Participants
Brief Title: A Study of LIPO-5 and ALVAC-HIV (vCP1452) as Possible HIV Vaccines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 042; ANRS VAC019; 10119 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2004-01-13; First posted 2004-01-14 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; ALVAC-HIV vCP1452; ALVAC Vaccine; HIV-1; Normal Values; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — ALVAC-HIV vCP1452

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- A (Experimental): Participants in Groups A will receive four injections over 6 months of either LIPO-5 or a placebo.
  Interventions: Biological: LIPO-5
- B (Experimental): Participants in Group B will receive four injections over 6 months of either the ALVAC-HIV (vCP1452) or a placebo.
  Interventions: Biological: ALVAC-HIV (vCP1452)
- C (Experimental): Participants in Groups C will receive six injections over 6 months. Participants in this group will receive either ALVAC-HIV (vCP1452) and LIPO-5 or a placebo. Participants who receive the vaccine combination will receive four injections of the same dose of ALVAC-HIV (vCP1452) and two injections of LIPO-5. The dose of LIPO-5 will be different for participants in Groups C, D, and E.
  Interventions: Biological: ALVAC-HIV (vCP1452); Biological: LIPO-5
- D (Experimental): Participants in Group D will receive six injections over 6 months. Participants in this group will receive either ALVAC-HIV (vCP1452) and LIPO-5 or a placebo. Participants who receive the vaccine combination will receive four injections of the same dose of ALVAC-HIV (vCP1452) and two injections of LIPO-5. The dose of LIPO-5 will be different for participants in Groups C, D, and E.
  Interventions: Biological: ALVAC-HIV (vCP1452); Biological: LIPO-5
- E (Experimental): Participants in Group E will receive six injections over 6 months. Participants in this group will receive either ALVAC-HIV (vCP1452) and LIPO-5 or a placebo. Participants who receive the vaccine combination will receive four injections of the same dose of ALVAC-HIV (vCP1452) and two injections of LIPO-5. The dose of LIPO-5 will be different for participants in Groups C, D, and E.
  Interventions: Biological: ALVAC-HIV (vCP1452); Biological: LIPO-5

INTERVENTIONS:
Biological: ALVAC-HIV (vCP1452) — experimental vaccine
  Arms: B; C; D; E
Biological: LIPO-5 — experimental vaccine
  Arms: A; C; D; E

SUMMARY:
This study will test the immune system response to and safety of two HIV vaccines alone and in combination: ALVAC-HIV (vCP1452) and LIPO-5. ALVAC-HIV (vCP1452) uses a canarypox virus with man-made parts of HIV attached to it. The canarypox virus cannot cause disease in people. LIPO-5 is a mixture of five man-made proteins similar to proteins found in HIV.

These vaccines are not produced from live HIV or from infected cells and do not contain the virus. It is not possible to become infected with HIV from these vaccines.

DETAILED DESCRIPTION:
Immune priming of cytotoxic T lymphocytes (CTLs) has been most successfully achieved with live attenuated virus or live virus vector vaccines. Recombinant canarypox vaccines have an excellent safety record and have induced HIV neutralizing antibodies and CTLs in early clinical trials. This study will evaluate the use of HIV lipopeptides (LIPO-5) alone and in combination with a canarypox-based HIV vaccine [ALVAC-HIV (vCP1452)] to further increase CTL activity.

Participants in this study will be randomly assigned to one of five groups. Participants in Groups A and B will receive four injections over 6 months. Participants in Group A will receive four injections of either LIPO-5 or a placebo. Participants in Group B will receive four injections of either the ALVAC-HIV (vCP1452) or a placebo. Participants in Groups C, D, and E will receive six injections over 6 months. Participants in these groups will receive either ALVAC-HIV (vCP1452) and LIPO-5 or a placebo. Participants who receive the vaccine combination will receive four injections of the same dose of ALVAC-HIV (vCP1452) and two injections of LIPO-5. The dose of LIPO-5 will be different for participants in Groups C, D, and E.

Participants will have 11 study visits over 18 months; the total duration of the study will be 30 months. The length of visits will vary and may last up to 3 hours. Study visits will include a medical interview, brief physical exam, and blood and urine tests. Participants will be tested for HIV before entering the study and at least five times during the study. All vaccine and placebo injections will be given in the upper arm muscle.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Willing to receive HIV test results
* Good general health
* Acceptable methods of contraception for females of reproductive potential
* Access to participating site and available for follow-up during the study

Exclusion Criteria:

* HIV vaccines or placebos in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first study vaccine administration
* Blood products within 120 days prior to first study vaccine administration
* Immunoglobulin within 60 days prior to first study vaccine administration
* Live attenuated vaccines within 30 days prior to first study vaccine administration
* Investigational research agents within 30 days prior to first study vaccine administration
* Subunit or killed vaccines within 14 days prior to first study vaccine administration
* Current tuberculosis prophylaxis or therapy
* Hypersensitivity to neomycin or egg products
* Uveitis, chronic Lyme disease, active mycobacterial diseases, or sarcoidosis
* Serious adverse reaction to a vaccine. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis
* Unstable asthma
* Type 1 or Type 2 diabetes mellitus
* Thyroid disease requiring treatment in the past 12 months
* Serious angioedema within the past 3 years
* Uncontrolled hypertension
* Bleeding disorder
* Malignancy unless it has been surgically removed and, in the opinion of the investigator, is not likely to recur during the study period
* Seizure disorder requiring medication within the past 3 years
* Asplenia
* Mental illness that would interfere with compliance with the protocol
* Other conditions that, in the judgment of the investigator, would interfere with the study
* Pregnant or breast-feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2004-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Immune response to vaccines | Throughout study
Clinical and laboratory adverse events | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Frey, Study Chair — St. Louis University; Larry Peiperl, Study Chair — San Francisco Dept. of Public Health
Locations (11):
- United States (11):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - Johns Hopkins Bloomberg School of Public Health,Ctr for Immunization Research,Project SAVE-Baltimore, Baltimore, Maryland
  - Project Brave HIV Vaccine CRS, Baltimore, Maryland
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - Fenway Community Health Clinical Research Site (FCHCRS), Boston, Massachusetts
  - Saint Louis Univ. School of Medicine, HVTU, St Louis, Missouri
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - NY Blood Ctr./Bronx CRS, The Bronx, New York
  - Miriam Hospital's HVTU, Providence, Rhode Island
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - FHCRC/UW Vaccine CRS, Seattle, Washington

REFERENCES:
- [Background] Evans TG, Keefer MC, Weinhold KJ, Wolff M, Montefiori D, Gorse GJ, Graham BS, McElrath MJ, Clements-Mann ML, Mulligan MJ, Fast P, Walker MC, Excler JL, Duliege AM, Tartaglia J. A canarypox vaccine expressing multiple human immunodeficiency virus type 1 genes given alone or with rgp120 elicits broad and durable CD8+ cytotoxic T lymphocyte responses in seronegative volunteers. J Infect Dis. 1999 Aug;180(2):290-8. doi: 10.1086/314895. PMID 10395842
- [Background] Klinguer C, David D, Kouach M, Wieruszeski JM, Tartar A, Marzin D, Levy JP, Gras-Masse H. Characterization of a multi-lipopeptides mixture used as an HIV-1 vaccine candidate. Vaccine. 1999 Sep;18(3-4):259-67. doi: 10.1016/s0264-410x(99)00196-6. PMID 10506650
- [Background] Pialoux G, Gahery-Segard H, Sermet S, Poncelet H, Fournier S, Gerard L, Tartar A, Gras-Masse H, Levy JP, Guillet JG; ANRS VAC 04 Study Team. Lipopeptides induce cell-mediated anti-HIV immune responses in seronegative volunteers. AIDS. 2001 Jul 6;15(10):1239-49. doi: 10.1097/00002030-200107060-00005. PMID 11426068
- [Background] Gahery-Segard H, Pialoux G, Figueiredo S, Igea C, Surenaud M, Gaston J, Gras-Masse H, Levy JP, Guillet JG. Long-term specific immune responses induced in humans by a human immunodeficiency virus type 1 lipopeptide vaccine: characterization of CD8+-T-cell epitopes recognized. J Virol. 2003 Oct;77(20):11220-31. doi: 10.1128/jvi.77.20.11220-11231.2003. PMID 14512570
- [Derived] Frey SE, Peiperl L, McElrath MJ, Kalams S, Goepfert PA, Keefer MC, Baden LR, Lally MA, Mayer K, Blattner WA, Harro CD, Hammer SM, Gorse GJ, Hural J, Tomaras GD, Levy Y, Gilbert P, deCamp A, Russell ND, Elizaga M, Allen M, Corey L. Phase I/II randomized trial of safety and immunogenicity of LIPO-5 alone, ALVAC-HIV (vCP1452) alone, and ALVAC-HIV (vCP1452) prime/LIPO-5 boost in healthy, HIV-1-uninfected adult participants. Clin Vaccine Immunol. 2014 Nov;21(11):1589-99. doi: 10.1128/CVI.00450-14. Epub 2014 Sep 24. PMID 25253665